CLINICAL TRIAL: NCT06386354
Title: Residual Neuromuscular Block in the Post-Anesthetic Unit and Postoperative Complications
Acronym: Porcerito
Status: Recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra-Bolaños, MD PhD, PhD, Dr. Negrin University Hospital
Other Study IDs: 2023-464-1
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Neuromuscular Block; Postoperative Complications
Keywords: General Anesthesia; Neuromuscular block
MeSH Terms: conditions — Postoperative Complications | interventions — Neuromuscular Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients submitted to General Anesthesia with Neuromuscular Block: Patients submitted to General Anesthesia with Neuromuscular Block
  Interventions: Diagnostic Test: Train-of-four

INTERVENTIONS:
Diagnostic Test: Train-of-four — Patients submitted to general anesthesia with neuromuscular block will be monitored at their arrival to the Post-Anesthesia Care Unit to assess the presence of residual neuromuscular block.

SUMMARY:
The use of neuromuscular blockers (NMB) is essential to optimize surgical conditions, ensure patient immobility during the intervention and prevent complications derived from involuntary movements. Intraoperative monitoring of neuromuscular relaxation allows the depth of neuromuscular blockade to be accurately evaluated, guaranteeing ideal conditions for the surgical team. Residual neuromuscular blockade (RNMB) is the persistence of muscle paralysis after the administration of NMB during a surgical intervention. The appearance of RNMB poses substantial challenges in the postoperative period, as it has negative repercussions for the safety and well-being of the patient.

DETAILED DESCRIPTION:
The use of neuromuscular blockers (NMB) is essential to optimize surgical conditions, ensure patient immobility during the intervention and prevent complications derived from involuntary movements. Intraoperative monitoring of neuromuscular relaxation allows the depth of neuromuscular blockade to be accurately evaluated, guaranteeing ideal conditions for the surgical team. Residual neuromuscular blockade (RNMB) is the persistence of muscle paralysis after the administration of NMB during a surgical intervention. The appearance of RNMB poses substantial challenges in the postoperative period, as it has negative repercussions for the safety and well-being of the patient. In this prospective observational study, all patients who underwent general anesthesia with neuromuscular blockade were studied consecutively to evaluate the presence of residual neuromuscular blockade and its potential consequences during hospital admission.Considering that the percentage of residual curarization is 19% (PORCzero study), with a 95% confidence interval and a 3% error margin, 236 patients are needed to accurately estimate the prevalence of residual curarization in the study population. With an expected loss proportion of 20%, the chosen sample size is 296 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing surgical intervention under general anesthesia that requires the use of neuromuscular block during the study time and that required hospital admission.
* Informed consent signature.

Exclusion Criteria:

* Neuromuscular disease
* Not having received neuromuscular block during the intervention
* Admission to the outpatient surgery unit
* Admission to the postoperative intensive care unit
* Patients who signed informed consent, but postoperative data could not be collected upon arrival at the PACU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical intervention under general anesthesia that requires the use of neuromuscular block during the study time.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Residual Neuromuscular Block | 5 minutes postoperatively
  Train-Of-Four ratio at arrival to the Post-Anesthetic Care Unit
Residual Neuromuscular Block | 8 minutes postoperatively
  Train-Of-Four ratio 3 minutes after the arrival to the Post-Anesthetic Care Unit

SECONDARY OUTCOMES:
Postoperative complications | 30 days postoperatively
  Postoperative complications during hospital admission

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Ángel Becerra, Las Palmas de Gran Canaria, Las Palmas

IPD SHARING:
Plan to Share IPD: Undecided